CLINICAL TRIAL: NCT00161356
Title: Blood, Bile and Tissue Pharmacokinetics of Single Dose Liposomal Amphotericin B (AmBisome ®) in Liver Transplant Patients.
Brief Title: Ambisome in Liver Transplant Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Budget issues
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Dr. Hadar Merhav, Memorial Hermann Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-04-0347; Astellas Pharma; APUSprojectno.JK-04-001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ambisome — 5mg/kg IV - one time dose during liver transplant
Procedure: Liver Biopsy — post drug delivery (60 min. after completion of Ambisome infusion)

SUMMARY:
In this study we are trying to find out the amount of a drug called Ambisome in the liver, the blood, the bile and the fatty tissues of the body. This drug is approved for treatment of infections caused by fungus and is known to be effective against most of the fungal infections, which can happen after liver transplantation. By taking small pieces (less than quarter of a teaspoon) of liver and fat during the liver transplant operation, we can measure how much of the drug is concentrated in the liver. After that, we will measure the level of the drug in the blood and in the bile that comes out of a small tube which is inserted into the bile tube as a routine in all liver transplant patients. These measurements will be taken daily for a week and then weekly for another 3 weeks.

We are inviting you to take part in this study in order to increase our knowledge of the behavior of this drug so that we can find the most effective treatment to prevent fungal infections in liver transplant patients.

DETAILED DESCRIPTION:
Fungal infections continue to be a source of serious morbidity and mortality in liver transplant patients. Liposomal Amphotericin B (AmBisome ®) has been shown in animals to be concentrated in the liver, lungs and leukocytes. It also has a long half-like making it a potentially attractive drug for prophylaxis in liver transplantation (OLT).

We propose to administer a single (5mg/kg) dose of AmBisome ® following reperfusion of the new liver. Liver, subcutaneous fat, blood and bile samples will be analyzed for AMB levels 1-2 hours after drug administration. Blood and bile, and body fluid samples will be sequentially analyzed for 3 weeks post transplant. This will be done in 50 consecutive patients. The incidence of fungal infections and adverse effects will be monitored for three months.

Persistent AMB levels in blood bile and ascites, if found, will provide a good rationale for AmBisome ® prophylaxis for fungal infections in outpatients.

ELIGIBILITY:
Inclusion Criteria:

* All adult liver transplant recipients receiving cadaveric liver transplants

Exclusion Criteria:

* Patients with choledocho-jejunostomy reconstruction of the biliary tree.
* Children less than 18 years of age
* Patients with known allergy to Amphotericin B.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Tissue concentration of ambisome | 3 months
Bile levels of amphotericin B over time (3 weeks) | 3 weeks
Blood levels of amphotericin B over time (3 weeks) | 3 weeks

SECONDARY OUTCOMES:
Rate of fungal infections | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hadar J. Merhav, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States